CLINICAL TRIAL: NCT01432041
Title: Brief Child Safety Interventions in Emergency Departments (Safety in Seconds)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Purpose: Prevention
Other Study IDs: JHSPH-H.31.02.04.03.B2
Record Dates: First submitted 2011-09-08; First posted 2011-09-12 (Estimated); Last update posted 2023-03-22 (Actual); Status verified 2011-09

CONDITIONS: Injury Prevention
Keywords: Injury prevention; smoke alarms; car seats

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: tailored health education — Health Information via a computer kiosk in the pediatric emergency department
  Other Names: Tailored health Communication

SUMMARY:
Safety in seconds is a randomized controlled trial of a computer tailored Injury Prevention program which was conducted in the waiting area of a level 1 pediatric trauma center. A computer kiosk was used to randomly assign participants to study groups, collect baseline data and generate tailored reports based on responses to assessment items. An intervention group received a personalized and stage-tailored safety report and a control group received a personalized, but otherwise generic report on other child health topics. Telephone follow-up interviews were conducted 2-4 weeks and again 4-6 months after enrollment. Home visits were completed for a subset (n=100) of parents who completed the 4-6 month follow-up interview. The study aimed to increase knowledge, self reported and observed safety behaviors.

ELIGIBILITY:
Inclusion Criteria:

* Eligible parents or guardians had to be English-speaking;
* have a child between 4-66 months of age seeking treatment for an injury or medical complaint, or have an age-appropriate sibling of a child being seen for these reasons;
* live in Baltimore City;
* and live with the child at least some of the time.

Exclusion Criteria:

-parents which did not meet inclusion criteria

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 901 (Actual)
Dates: Start 2004-09; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Knowledge outcome
  Measures of Home safety Knowledge
Reported and Observed Home Safety behaviors
  Reportedf and Observed Home Safety Behaviors (Car Seats, Smoke Alarms)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea C Gielen, ScD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health

REFERENCES:
- [Background] Gielen AC, McKenzie LB, McDonald EM, Shields WC, Wang MC, Cheng YJ, Weaver NL, Walker AR. Using a computer kiosk to promote child safety: results of a randomized, controlled trial in an urban pediatric emergency department. Pediatrics. 2007 Aug;120(2):330-9. doi: 10.1542/peds.2006-2703. PMID 17671059